CLINICAL TRIAL: NCT04155190
Title: A Multicenter, Randomized, Double Blind, Vehicle-controlled, Phase 2 Efficacy and Safety Study of Patidegib Topical Gel, 2%, for the Reduction of Disease Burden of Persistently Developing Basal Cell Carcinomas (BCCs) in Patients With Non-Gorlin High Frequency BCC
Brief Title: An Study of Patidegib Topical Gel, 2%, for the Reduction of Disease Burden of Persistently Developing Basal Cell Carcinomas in Patients With Non-Gorlin High Frequency BCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to low blinded event rate
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pelle-926-203
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Basal Cell Carcinoma
Keywords: High Frequency Basal Cell Carcinoma; non-gorlin; HF-BCC; Bazex-Dupré-Christol Syndrome; Rombo Syndrome; Oley Syndrome; Xeroderma Pigmentosum (XP) Syndrome; BCC; SEB; Hedgehog inhibitor; Basal Cell Nevus Syndrome; Basal Cell Carcinoma; Surgically Eligible Basal Cell Carcinoma; patidegib; HFBCC; HHI
MeSH Terms: conditions — Carcinoma, Basal Cell; Rombo syndrome; Xeroderma Pigmentosum; Syndrome; Basal Cell Nevus Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) to receive either Patidegib Topical Gel, 2%, or Vehicle for 9 months. Randomization will be stratified by gender.
Who Masked: Participant, Care Provider, Investigator
Masking Description: As a double-blinded study, the Investigators, the site staff, PellePharm, and the Clinical Monitor(s) will be blinded to the treatment assigned to individual subjects. Delegated staff members at the study site will dispense the investigational product (IP) and will collect and weigh all used and unused IP tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patidegib Topical Gel, 2% (Experimental): Participants will be randomized (1:1) to receive Patidegib Topical Gel, 2% for 9 months
  Interventions: Drug: Patidegib Topical Gel, 2%
- Patidegib Topical Gel, Vehicle (Active Comparator): Participants will be randomized (1:1) to receive Patidegib Topical Gel, Vehicle for 9 months
  Interventions: Drug: Patidegib Topical Gel, Vehicle

INTERVENTIONS:
Drug: Patidegib Topical Gel, 2% — Patidegib Topical Gel, 2%
  Other Names: IP
  Arms: Patidegib Topical Gel, 2%
Drug: Patidegib Topical Gel, Vehicle — Patidegib Topical Gel, Vehicle
  Other Names: IP, Vehicle
  Arms: Patidegib Topical Gel, Vehicle

SUMMARY:
This is a multicenter, randomized, double-blind, stratified, vehicle-controlled study of the efficacy and safety of Patidegib Topical Gel, 2%, applied topically twice daily to the face of adult participants with non-Gorlin HF-BCC (high-frequency basal cell carcinoma). Participants will be randomized (1:1) to receive either Patidegib Topical Gel, 2%, or Vehicle for 9 months. Randomization will be stratified by gender. The primary endpoint is the number of nSEB (surgically eligible basal cell carcinoma) that develop on the face over the 9 month period. The primary end point will be assessed by imaging and tracking of BCCs consistently throughout the study in order to identify nSEBs.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have had at least 10 (with at least 3 on the face) clinically typical BCCs present within 24 months prior to Screening and Randomization (Baseline/Day 1). Additionally, the subject must have at least 2 BCCs with longest diameter <5 mm present on the face prior to Screening and Randomization (Baseline/Day 1).
2. The subject must be willing to abstain from application of a non-study topical medication (prescription or over the counter) to facial skin for the duration of the trial except as prescribed by the Investigator.

Exclusion Criteria:

1. The subject has been previously diagnosed with Gorlin syndrome
2. On medical history, family history or clinical examination there is a suspicion that the patient has Gorlin syndrome.
3. Patients with a family history of medulloblastoma
4. The subject has used topical treatment to the face or systemic therapies that might interfere with the evaluation of the study IP.
5. The subject has uncontrolled systemic disease.
6. The subject has been treated for invasive cancer within the past 5 years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or chronic lymphocytic leukemia (CLL) Stage 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Number of new surgically eligible BCCs (nSEBs) | Baseline through Month 9

SECONDARY OUTCOMES:
Number of treatment emergent adverse events assessed with means and standard errors or proportions | Baseline through Month 9

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Operations, Study Director — PellePharm, Inc.
Locations (14):
- United States (14):
  - Axiom Research, LLC, Apple Valley, California
  - Axiom Research, LLC, Colton, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - The Dermatology Center of Newport, Newport Beach, California
  - Palm Beach Dermatology Research, Delray Beach, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - PellePharm Investigative Site, Saint Augustine, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Grekin Skin Institute, Warren, Michigan
  - PellePharm Investigative Site, Henderson, Nevada
  - Skin Laser and Surgery Specialists of NY&NJ, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University of Utah, Murray, Utah

IPD SHARING:
Plan to Share IPD: Undecided